CLINICAL TRIAL: NCT03851731
Title: Pharmacokinetic Evaluation of Intranasal Naltrexone and Naloxone Administered Separately and in Combination in Healthy Volunteers
Brief Title: Evaluation of Intranasal Naltrexone and Naloxone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Naltrexone-Ph1a-001
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2019-02

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; vivitrol; Naloxone; 6 beta-hydroxynaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Naltrexone (Experimental): Subject received a single intranasal dose of 2 mg naltrexone for a total of 3 times in a 13 day period with a 4-day washout period between each does until all treatments were administered
  Interventions: Drug: Naltrexone
- Naloxone (Experimental): Subject received a single intranasal dose of 4 mg naloxone for a total of 3 times in a 13 day period with a 4-day washout period between each does until all treatments were administered
  Interventions: Drug: Naloxone
- Naltrexol (Experimental): Subject received a single intranasal dose of a combination of 2 mg naltrexone and 4 mg naloxone for a total of 3 times in a 13 day period with a 4-day washout period between each does until all treatments were administered
  Interventions: Drug: Naltrexol

INTERVENTIONS:
Drug: Naltrexone — Intranasal spray
  Other Names: Vivitrol
  Arms: Naltrexone
Drug: Naloxone — Intranasal spray
  Other Names: Narcan
  Arms: Naloxone
Drug: Naltrexol — Intranasal spray
  Arms: Naltrexol

SUMMARY:
This study will be to determine the pharmacokinetics of naltrexone and naloxone when administered via intranasal separately and in combination in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 55 years of age, inclusive.
* Provide written informed consent.
* Body mass index (BMI) ranging from 18 to 30 kg/m2, inclusive.
* Adequate venous access.
* No clinically significant concurrent medical conditions determined by medical history, physical examination, clinical laboratory examination, vital signs, and 12-lead ECG.
* Agree to use a reliable double-barrier method of birth control from the start of screening until one week after completing the study. Oral contraceptives are prohibited.
* Agree not to ingest alcohol, drinks containing xanthine >500 mg/day (e.g., Coca Cola®, tea, coffee, etc.), or grapefruit/grapefruit juice or participate in strenuous exercise 72 hours prior to admission through the last blood draw of the study.

Exclusion Criteria:

* Contact site for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2015-11-07 (Actual); Study Completion 2015-11-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter [maximum serum concentration - Cmax] | 12 days
  The primary endpoints of the study are the pharmacokinetic parameter, maximum serum concentration [Cmax], of naltrexone and naloxone when administered and in combination.
Pharmacokinetic parameter [area under the plasma concentration time curve - AUCO-t] | 12 days
  The primary endpoints of the study are the pharmacokinetic parameter, area under the plasma concentration time curve [AUCO-t] of naltrexone and naloxone when administered and in combination.
Pharmacokinetic parameter [area under the plasma concentration curve from zero to infinity - AUCO-inf] | 12 days
  The primary endpoints of the study are the pharmacokinetic parameter, area under the plasma concentration curve from zero to infinity [AUCO-inf] of naltrexone and naloxone when administered and in combination.

SECONDARY OUTCOMES:
Adverse Events | 15 days
  To assess and document any adverse events measures
Vital Sign - Heart Rate | 12 days
  To assess and document heart rate before and after intranasal dosing
Vital Sign - Blood pressure (diastolic) | 12 days
  To assess and document blood pressure (diastolic) before and after intranasal dosing
Vital Sign - Blood pressure (systolic) | 12 days
  To assess and document blood pressure (systolic) before and after intranasal dosing
Vital Sign - Respiration Rate | 12 days
  To assess and document respiration rate before and after intranasal dosing
Electrocardiogram | 12 days
  Twelve-lead ECGs performed according to standard procedures that will assess P wave, PR interval, QRS complex, ST segment, T wave and QT interval.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Chiang, PhD, Study Chair — NIH / NIDA

IPD SHARING:
Plan to Share IPD: No